CLINICAL TRIAL: NCT03221530
Title: Early Intervention for Suicide Risk Among Immigrant Youth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kiara Alvarez, Instructor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017P001429
Record Dates: First submitted 2017-07-16; First posted 2017-07-18 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Family Conflict; Suicidal Ideation
Keywords: suicidal ideation; mental health; adolescent; Latino; immigrant
MeSH Terms: conditions — Suicidal Ideation; Psychological Well-Being | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EISR-I (Experimental): Participants in the Early Intervention for Suicide Risk Among Immigrant Youth (EISR-I) family-based intervention will attend 8 in-person sessions with at least one parent/guardian.
  Interventions: Behavioral: Early Intervention for Suicide Risk Among Immigrant Youth
- Enhanced usual care (Active Comparator): Participants in the usual care arm will receive a safety planning and assessment feedback session from the research team and will receive usual care in the behavioral health clinic where the study takes place.
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Early Intervention for Suicide Risk Among Immigrant Youth — The EISR-I intervention includes family treatment engagement, shared problem definition, and sessions designed to address family cohesion, communication, and conflict resolution.
  Arms: EISR-I
Behavioral: Enhanced usual care — This intervention includes a session with the family to engage in safety planning and provide feedback on their baseline assessment data.
  Arms: Enhanced usual care

SUMMARY:
The purpose of this project is to develop and test a family-based preventive intervention for suicide risk among 1st and 2nd generation immigrant Latino/a adolescents. The intervention will focus on reducing suicide risk by reducing family conflict and intergenerational cultural conflict and improving parent-child communication. The investigators will first develop the 8-session preventive intervention with quantitative data from analysis of existing longitudinal studies and qualitative feedback from Latino youth and their caregivers, clinicians, administrators, and research consultants, as well as results from initial pilot testing of the intervention. The investigators will then conduct a pilot randomized trial with 40 adolescents and their families to test feasibility, acceptability, and impact on intervention targets. Successful development of the intervention would improve mental health outcomes for a growing and underserved portion of the U.S. population.

DETAILED DESCRIPTION:
Suicide is the second-leading cause of death among adolescents, with rates increasing between 1999 and 2014. Family-based preventive interventions demonstrate promise for reducing suicide risk among adolescents, and are particularly relevant for addressing suicide risk factors specific to immigrant youth, who comprise one-fourth of the U.S. population under 18. The purpose of this project is to develop and test a family-based preventive intervention for suicide risk among 1st and 2nd generation immigrant Latino/a adolescents. In the first phase of intervention development, quantitative and qualitative data will be used to develop and if necessary refine a new family based preventive intervention (Early Intervention for Suicide Risk among Immigrant Youth, EISR-I). The investigators will then test the intervention in a pilot case series in order to finalize assessment and intervention protocols. In the second phase, the investigators will pilot test the preventive intervention, delivered by mental health clinicians to 1st and 2nd generation Latino/a early adolescents and their families, in order to assess feasibility, acceptability, and impact on the intervention targets (i.e. a positive signal of the intervention) on the study population. Twenty families will be randomized to receive the 8-session intervention and twenty will receive enhanced usual care including a safety planning and feedback session.

ELIGIBILITY:
Inclusion Criteria:

* Latino
* First generation (foreign-born) or second-generation (at least one parent foreign-born) immigrant
* 12 to 15 years old
* Speaks English or Spanish
* Reports current suicidal ideation with no plan, past-year suicidal ideation, or a suicide plan more than three months prior OR has a CAT-SS score>34

Exclusion Criteria:

* Suicide attempt in the past three months
* Endorses psychotic symptoms on a pre-study screener
* Has severe major depressive disorder
* Has a prior diagnosis of severe intellectual disability
* Receiving individual or family therapy

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Columbia Suicide Severity Rating Scale Screener (C-SSRS); change from baseline at multiple time points | baseline, 3, 6, and 12 months
  A self-report scale of suicidal ideation, plans and attempts

SECONDARY OUTCOMES:
Computerized Adaptive Test - Suicide Scale (CAT-SS); change from baseline at multiple time points | baseline, 3, 6, and 12 months
  A computerized adaptive suicide scale that provides a continuous self-report measure of suicide risk
Family Relationship Index; change from baseline at multiple time points | baseline, 3, 6, and 12 months
  A self-report measure that provides an overall index of the quality of the family environment, as well as subscores that reflect family cohesion, expressiveness, and conflict.
Family Cultural Conflict Scale; change from baseline at multiple time points | baseline, 3, 6, and 12 months
  A self-report measure of conflicts within a family related to cultural values and practices.
Parent-Adolescent Communication Scale; change from baseline at multiple time points | baseline, 3, 6, and 12 months
  A self-report measure of the quality of communication between adolescent and parent.

IPD SHARING:
Plan to Share IPD: No